CLINICAL TRIAL: NCT00771459
Title: Lokal Infiltrations Analgesi Med Ropivakain 0,5 % Versus Placebo Ved Rygkirurgi for Spinalstenose: et Prospektivt Randomiseret, Dobbeltblindet, Placebo-kontrolleret Studie
Brief Title: Local Infiltration Analgesia in Major Spine Surgery With Ropivacaine Versus Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Billy B Kristensen, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-D-2007-0111
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2008-10

CONDITIONS: Pain, Postoperative
Keywords: Local infiltration analgesia; postoperative pain; ropivacaine
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Ropivacaine (Active Comparator)
  Interventions: Drug: Ropivacaine 0.5 %
- Placebo (Placebo Comparator)
  Interventions: Drug: Isotonic NaCl

INTERVENTIONS:
Drug: Ropivacaine 0.5 % — Local infiltration analgesia
  Arms: Ropivacaine
Drug: Isotonic NaCl — Local infiltration analgesia
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine whether local infiltration analgesia (LIA) with Ropivacaine and adrenaline is effective in the treatment of postoperative pain after major spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients eligible for major spine surgery
* must speak and understand Danish
* must be able to give oral and written consent

Exclusion Criteria:

* alcohol or medicine abuse
* treatment with opioids > 100 mg daily
* allergy to local anesthetics
* severe obesity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | 0-48 h postoperatively

SECONDARY OUTCOMES:
Analgesia consumption | 0-48 h postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark